CLINICAL TRIAL: NCT03869749
Title: Decreasing Stress and Anxiety in Adolescents From High-Conflict Homes: Testing a Mindfulness Group + Ecological Momentary Intervention
Brief Title: The Moving 2 Mindful (M2M) Study: Mindfulness Group + Ecological Momentary Intervention
Acronym: M2M
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped early due to lack of enrollment.
Sponsor: Colorado State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2M; K01AT009592 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-03-11 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders | interventions — Health

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two study interventions in an open randomized trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The majority of study personnel, including the PI and study statistician, will be blinded until database lock. All individuals who will be involved with endpoint assessment will be blinded until database lock. Intervention facilitators will not be blinded, but will not be involved in endpoint assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learning to BREATHE Plus (Experimental): It is a 6-week manualized program; each meeting is 1.5 hours, for a total of 9 contact hours. It will be administered in a classroom at Colorado State University. Adolescents will be sent ecological momentary intervention text messages several times a day (with reminders, encouragement, and guides to practice mindfulness), and also have access to an on demand online library of mindfulness resources.
  Interventions: Behavioral: Learning to BREATHE Plus
- Health and wellness (Active Comparator): It is a 6-week program; each meeting is 1.5 hours, for a total of 9 contact hours. It will be administered in a classroom at Colorado State University.
  Interventions: Behavioral: Health and wellness

INTERVENTIONS:
Behavioral: Learning to BREATHE Plus — Activities include psycho-education about stress and emotion regulation, and practices of body scanning, non-aerobic yoga, and meditation, which are designed to cultivate and provide opportunities to practice present-focused, non-judgmental attention.
  Arms: Learning to BREATHE Plus
Behavioral: Health and wellness — The Health Education Wellness Program (modeled after Hey Durham) (Bravender, 2005) will provide didactic information on substance use, nutrition/body image, stress management, exercise, and signs of depression/suicide.
  Arms: Health and wellness

SUMMARY:
This study will evaluate the feasibility and acceptability of Learning to BREATHE (a mindfulness intervention for adolescents) plus an ecological momentary intervention (Learning to Breathe Plus), and will examine the extent to which mindfulness reduces dysregulated stress physiology, perceived stress, and anxiety in adolescents from high conflict homes.

DETAILED DESCRIPTION:
Adolescents from homes with interparental conflict will be randomly assigned to Learning to BREATHE Plus (the standard group program designed to increase mindfulness, plus a multi-method adaptive intervention that will be comprised of an ecological momentary intervention and online library of mindfulness practices) or to a health and wellness active control condition to determine feasibility, acceptability, and potential effectiveness of Learning to BREATHE Plus.

ELIGIBILITY:
Inclusion Criteria:

* two parents in the home
* an adolescent who is between 14 and 18 years of age
* marital distress and/or problematic interparental conflict (based on parent or youth reports)
* youth reports of stress or anxiety

Exclusion Criteria:

* two parents in the home, but they are pursuing legal divorce or separation
* parents are not willing to receive marital education/support
* adolescents are severely clinically depressed or report suicidal ideation at baseline

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Safe implementation | Across 8-week intervention period
  Implementation without increase in symptomatology
Recruitment of target sample size | Across 8-week intervention period
  Successful recruitment of 38 families (114 individuals)
Enrollment of percent eligible | Across 8-week intervention period
  Enrolling a high percent of eligible families to the study/intervention
Retention to interventions | Across 8-week intervention period
  A high proportion of adolescents will attend 4/6 sessions

SECONDARY OUTCOMES:
Feasibility of implementation | Across 8-week intervention period
  Successful implementation and retention to study (i.e., fidelity of intervention delivery >=80%, <=5% reports of not receiving ecological momentary intervention from adolescents, >=90% attendance at 4/6 sessions, >= retainment at post-group and follow-up)
Acceptability of interventions | Across 8-week intervention period
  Rated by participants

OTHER OUTCOMES:
Mindfulness, self-reported | Up to 3 months of follow-up
  Adolescents reported mindfulness (Mindfulness Awareness and Attention Scale, Adolescent Version; Brown, West, Loverich, & Biegel, 2011). There are 14 items on this scale, each answered on a scale from 1 (almost always) to 6 (almost never). Answer across 14 items are averaged such that higher scores indicate higher trait mindfulness (minimum = 1; maximum = 6).
Mindfulness, observed | Up to 3 months of follow-up
  Adolescents observed distress tolerance, an important component of mindfulness (Behavioral Indicator of Resiliency to Distress; Lejeuz et al., 2006)
Self-compassion, self-reported | Up to 3 months of follow-up
  Self-Compassion Scale, short form (Raes, Pommier, Neff, & Van Gucht, 2011). This scale has 12 items, answered on a scale from 1 (almost never) to 5 (almost always). There are 6 subscales measured on this scale, each with 2 items: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Subscale and total scores are calculated based on means after reverse scoring so that high scores indicate higher self-compassion (minimum: 1; maximum: 5).
Adolescent reports of emotion regulation | Up to 3 months of follow-up
  Emotion regulation (Difficulties in Emotion Regulation Scale; Gratz & Roemer, 2004). This scale has 36 items that measure difficulties in 6 sub-dimensions of emotion regulation: nonacceptance of emotional responses (6 items: minimum: 1; maximum: 36), difficulties engaging in goal-directed behavior (5 items: minimum: 1; maximum: 30), impulse control difficulties (6 items: minimum: 1; maximum: 36), lack of emotional awareness (6 items: minimum: 1; maximum: 36), limited access to emotion regulation strategies (8 items: minimum: 1, maximum 48), and lack of emotional clarity (5 items: minimum: 1; maximum: 30). Questions are answered on a scale from 1 (almost never) to 5 (almost always). Subscale and total scores are summed such that higher scores indicate greater difficulties with emotion regulation (total scores: minimum: 1, maximum: 180).
Anxiety | Up to 3 months of follow-up
  Parent and adolescent reported youth anxiety (Revised Child Anxiety and Depression Scale; Chorpita, Yim, Moffitt, Umemoto, & Francis, 2000). This scale has 47 items answered on a scale from 0 (never) to 3 (always), and answers are summed. Total scores range from 0 to 141, with higher scores reflecting more symptoms of anxiety and depression. Subscales can also be used to calculate scores for separation anxiety (7 items; minimum: 0, maximum: 21), social anxiety (9 items; minimum: 0, maximum 27), obsessive/compulsions (6 items; minimum: 0, maximum: 18), panic/agoraphobia (9 items; minimum: 0, maximum: 27), generalized anxiety (6 items; minimum: 0, maximum: 18), and major depression (10 items; minimum: 0, maximum: 30), with higher scores reflecting more symptoms.
Cortisol stress reactivity | Up to 3 months of follow-up
  Cortisol reactivity to a stressor (saliva samples after baseline and immediately as well as 10 and 20m after stressor); area under the curve will be calculated
Cardiovascular stress reactivity | Up to 3 months of follow-up
  Adolescent cardiovascular reactivity to a stressor (across three minutes intervals at baseline and during the stressor); change from baseline to stressor will be calculated
Diurnal cortisol production | Up to 3 months of follow-up
  Cortisol production across the day (participants will be asked to provide samples upon awakening, 30 minutes after waking, at 4:00 PM, and before brushing their teeth for bed) to calculate cortisol awakening responses and decreases in cortisol production from morning to evening

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Researchers interested in using these data to test novel hypotheses can contact the corresponding author and submit a data proposal form to be reviewed by the study team.

REFERENCES:
- [Background] Lucas-Thompson R, Seiter N, Broderick PC, Coatsworth JD, Henry KL, McKernan CJ, Smyth JM. Moving 2 Mindful (M2M) study protocol: testing a mindfulness group plus ecological momentary intervention to decrease stress and anxiety in adolescents from high-conflict homes with a mixed-method longitudinal design. BMJ Open. 2019 Nov 28;9(11):e030948. doi: 10.1136/bmjopen-2019-030948. PMID 31784436